CLINICAL TRIAL: NCT06975449
Title: Validation the Effectiveness of Graded Training in the MultiComponent Physical Exercise Program (Vivifrail) Among Senile Care Center Residents: A Randomized Controlled Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Shu Hua Lu, Associate Professor, China Medical University Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CMUH114-REC3-034
Record Dates: First submitted 2025-04-28; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Frailty; Physical Inactivity; Aging
MeSH Terms: conditions — Frailty; Sedentary Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group: Usual Care (Active Comparator): Participants in this group will receive usual care with no structured physical activity program. They will continue their normal daily routines and have access to health education materials unrelated to physical activity.
  Interventions: Behavioral: Multicomponent Physical Exercise Program (Vivifrail)
- Intervention Group: Multicomponent Physical Activity Program (Vivifrail) (Experimental): Participants in this arm will receive a 12-week multicomponent physical activity program based on the Vivifrail protocol, designed to improve physical function and reduce frailty in older adults. The intervention includes individualized exercise sessions incorporating strength, balance, flexibility, and endurance training, adjusted according to baseline functional capacity. Sessions are supervised by trained personnel and conducted three times per week in a community or long-term care setting. The program also includes educational components promoting adherence and safe exercise practices.
  Interventions: Behavioral: Multicomponent Physical Exercise Program (Vivifrail)

INTERVENTIONS:
Behavioral: Multicomponent Physical Exercise Program (Vivifrail) — Vivifrail physical training, 5 times/week, 50-60 minutes/session for 12 weeks

SUMMARY:
This study evaluates the effectiveness of the Vivifrail multicomponent physical exercise program among elderly residents with different levels of frailty in long-term care centers. A 12-week intervention will be conducted in randomly assigned experimental and control groups. Outcomes include physical performance, fall risk, grip strength, calf circumference, and ICOPE function.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥70, resident in LTC center, ambulatory, physician-cleared for training

Exclusion Criteria:

* Conditions listed in Vivifrail exclusion criteria (e.g., acute MI, unstable angina, recent fractures, uncontrolled hypertension, etc.)

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
SPPB Score change at Weeks 0, 4, 8, 12, 16, 20, 24 | SPPB Score change at Weeks 0, 4, 8, 12, 16, 20, 24
  SPPB Score change at Weeks 0, 4, 8, 12, 16, 20, 24
Fall risk assessment (TUG, gait speed, number of falls) at Weeks 0, 4, 8, 12, 16, 20, 24 | Fall risk assessment (TUG, gait speed, number of falls) at Weeks 0, 4, 8, 12, 16, 20, 24
  Fall risk assessment (TUG, gait speed, number of falls) at Weeks 0, 4, 8, 12, 16, 20, 24

SECONDARY OUTCOMES:
ICOPE function assessment at Weeks 0, 12, 24 | ICOPE function assessment at Weeks 0, 12, 24
  ICOPE function assessment at Weeks 0, 12, 24
Grip strength (hand dynamometer) at Weeks 0, 12, 24 | Grip strength (hand dynamometer) at Weeks 0, 12, 24
  Grip strength (hand dynamometer) at Weeks 0, 12, 24

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No